CLINICAL TRIAL: NCT06663449
Title: Comparison of ESP Block and STAP Plane Block in Laparoscopic Cholecystectomy Surgery
Brief Title: Comparison of ESP Block and STAP Plane Block
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Sevim Cesur, principal investigator, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KAEK/13.bI.04
Record Dates: First submitted 2024-10-14; First posted 2024-10-29 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Postoperative Pain
Keywords: regional anesthesia; Erector spinae plane block; subcostal transversus abdominis plane block
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP USING subcostal transversus abdominis plane block (Active Comparator): Before being taken to the surgical table preoperatively, monitoring and sedation will be performed in the operating room block unit, then subcostal tap block will be performed and postoperative PCA will be applied.Patients' perioperative pain will be monitored with a NOL (nociception level) monitor. The remifentanil dose will be adjusted to keep the NOL level between 10 and 25. After the patients are followed up for 24 hours postoperatively, their additional analgesia needs and amounts during this period will be compared.
  Interventions: Procedure: subcostal transversus abdominis plane block
- GROUP USING erector spinae plane block (Active Comparator): Before being taken to the surgical table preoperatively, monitoring and sedation will be performed in the operating room block unit, then erector spinae plane block will be performed and postoperative PCA will be applied.Patients' perioperative pain will be monitored with a NOL (nociception level) monitor. The remifentanil dose will be adjusted to keep the NOL level between 10 and 25. After the patients are followed up for 24 hours postoperatively, their additional analgesia needs and amounts during this period will be compared.
  Interventions: Procedure: erector spinae plane block

INTERVENTIONS:
Procedure: subcostal transversus abdominis plane block — subcostal transversus abdominis plane block will be performed using 20 mL of 0.25 bupivacaine
  Arms: GROUP USING subcostal transversus abdominis plane block
Procedure: erector spinae plane block — erector spinae plane block will be performed using 20 mL of 0.25 bupivacaine
  Arms: GROUP USING erector spinae plane block

SUMMARY:
In order to effectively manage postoperative analgesia in patients planned to undergo elective laparoscopic cholecystectomy, patients will be divided into 2 (two) groups and informed consent forms will be obtained after the necessary information is provided so that both groups can be included in the study. In the group planned to undergo erector spinae plane block, erector spinae plane block will be performed after monitoring and sedation in the operating room block unit before being taken to the surgical table preoperatively and postoperative PCA analgesia will be applied. In patients who will undergo subcostal transversus abdominis plane block, subcostal tap block will be performed after monitoring and sedation in the operating room block unit before being taken to the surgical table preoperatively and postoperative PCA analgesia will be applied. The patients' perioperative pain will be monitored with NOL (nociception level) monitor. Remifentanil dose will be adjusted to keep the NOL level between 10 and 25. After the patients are followed up for 24 hours postoperatively, their additional analgesia needs and amounts during this process will be compared. In this way, it is aimed to show that the analgesic method can be used effectively in the follow-up of pain management by comparing the Erector Spina Plane block and the Subcostal Transversus Abdominis Plane block as an effective analgesic application in laparoscopic cholecystectomy operations.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will undergo laparoscopic cholecystectomy:
* 18-75 years old
* ASA I-II-III patients

Exclusion Criteria:

* Use of anticoagulant drugs
* Known allergy to drugs to be used
* Infection in the area where the block will be performed
* Patient's reluctance

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2024-12-15 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
NRS Scores | 1 hours after surgery(T1), 3 hours after surgery (T2), 6 hours after surgery (T3), 12 hours after surgery (T4) and 24 hours after surgery(T5)
  NRS scores of the patients after the surgery (0=no pain, 10=worst pain imaginable)
Morphine consumption | 1 hours after surgery(T1), 3 hours after surgery (T2), 6 hours after surgery (T3), 12 hours after surgery (T4) and 24 hours after surgery(T5)
  Amount of morphine consumption (mg)

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli University, Kocaeli, Turkey (Türkiye)

REFERENCES:
- [Result] Hashemi SJ, Heydari SM, Hashemi ST. Paravertebral block using bupivacaine with/without fentanyl on postoperative pain after laparoscopic cholecystectomy: A double-blind, randomized, control trial. Adv Biomed Res. 2014 Sep 4;3:187. doi: 10.4103/2277-9175.140099. eCollection 2014. PMID 25250301
- [Result] Agarwal A, Batra RK, Chhabra A, Subramaniam R, Misra MC. The evaluation of efficacy and safety of paravertebral block for perioperative analgesia in patients undergoing laparoscopic cholecystectomy. Saudi J Anaesth. 2012 Oct-Dec;6(4):344-9. doi: 10.4103/1658-354X.105860. PMID 23493523
- [Result] Mimic A, Bantel C, Jovicic J, Mimic B, Kisic-Tepavcevic D, Durutovic O, Ladjevic N. Psychological factors as predictors of early postoperative pain after open nephrectomy. J Pain Res. 2018 May 9;11:955-966. doi: 10.2147/JPR.S152282. eCollection 2018. PMID 29785136
- [Result] Vrsajkov V, Ilic N, Uvelin A, Ilic R, Lukic-Sarkanovic M, Plecas-Duric A. Erector spinae plane block reduces pain after laparoscopic cholecystectomy. Anaesthesist. 2021 Dec;70(Suppl 1):48-52. doi: 10.1007/s00101-021-01015-5. Epub 2021 Oct 18. PMID 34661682
- [Result] Kim S, Bang S, Kwon W. Intermittent erector spinae plane block as a part of multimodal analgesia after open nephrectomy. Chin Med J (Engl). 2019 Jun 20;132(12):1507-1508. doi: 10.1097/CM9.0000000000000269. No abstract available. PMID 31205117
- [Result] Tulgar S, Selvi O, Kapakli MS. Erector Spinae Plane Block for Different Laparoscopic Abdominal Surgeries: Case Series. Case Rep Anesthesiol. 2018 Feb 18;2018:3947281. doi: 10.1155/2018/3947281. eCollection 2018. PMID 29670771
- [Result] Grass JA. Patient-controlled analgesia. Anesth Analg. 2005 Nov;101(5 Suppl):S44-S61. doi: 10.1213/01.ANE.0000177102.11682.20. PMID 16334492